CLINICAL TRIAL: NCT02120404
Title: Pilot Phase II Study: Hemodynamic Tolerance and Anti-inflammatory Effects of Esmolol During the Treatment of Septic Shock
Acronym: THANE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120912; 2013-005174-22 (EudraCT Number)
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Septic Shock
Keywords: septic shock, hemodynamic tolerance, esmolol
MeSH Terms: conditions — Shock, Septic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (GC) (No Intervention): Control group: no esmolol administration
- Group 10 (G10) (Experimental): Esmolol titrated in order to reduce heart rate by 10% as compared to baseline heart rate
  Interventions: Drug: Esmolol administration
- Group 20 (G20) (Experimental): Esmolol titrated in order to reduce heart rate by 20% as compared to baseline heart rate
  Interventions: Drug: Esmolol administration

INTERVENTIONS:
Drug: Esmolol administration — Esmolol will be administered during 24 hours, beginning with a titration period to determine the minimal dose allowing to achieve the randomized heart rate reduction of 10% or 20%, as defined by randomization.
  Titration will be performed in sequences of increasing doses, beginning with 5 μg/kg/min as initial dose, and increasing by 5 μg/kg/min each 30 minutes until the target heart rate reduction is obtained. The maximum dose is 200 μg/kg/min.
  The titrated dose will be maintained for a total duration of 24 hours.
  Other Names: BREVIBLOC 10 mg/ml
  Arms: Group 10 (G10); Group 20 (G20)

SUMMARY:
The purpose of this study is :

- to evaluate the hemodynamic tolerance of esmolol titrated to obtain a lowering of heart rate of 10% or 20%.

DETAILED DESCRIPTION:
During septic shock, the consequences of treatment by a β1-blocker on inflammation and cardiovascular variability are unknown. The use of esmolol should have positive effects on inflammation and hemodynamic tolerance. These effects are probably dose-dependent.

The study will enroll adult patients hospitalized in ICU, for severe septic shock requiring treatment by a vasopressor.

A total of 45 patients will be included. Among these 45 patients, 15 patients will be randomized in the control group. 30 patients will be randomized to Esmolol with the objective to decrease heart rate by 10% (Group G10, n=15) or 20% (Group G20, n=15). Esmolol will be administered for 24 hours.

This multicenter study will be performed in 3 investigation sites.

The following parameters will be evaluated at different moments during the 28 days follow up of each patient, mainly:

* Origin of sepsis, SOFA score.
* Hemodynamic parameters will be continuously recorded for the 24 hours of experimental period.
* Cardiovascular variability (arterial pressure and heart rate) will be recorded for 24 hours.
* 3 echocardiograms at H0, H12 and H24 will be performed.
* Biological parameters will be sampled at H0, H6, H12 and H24: They include standard biological parameters (Urea, Creatinin, Bilirubin,……) and specific parameters (catecholamines, vasopressin, insulin, cortisol, proinflammatory cytokines and anti-inflammatory cytokines. Dosages will be performed only at H0, H12 and H24 in order to study:

  * The expression of adrenergic receptors and their genetic polymorphisms on circulating immune cells.
  * The Th1/Th2 balance in immune cells.

Each patient will be followed-up for 28 days.

The variation of MAP and of cardiac output induced by esmolol should not exceed 15% of baseline values. If the variation is more important esmolol administration will be stopped and the hemodynamical tolerance will be defined as poor.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years;
* Patient with septic shock;
* Patient with arterial catheter, central venous catheter with PVC and PiCCO;
* Consent signed by patient. In the absence of a consent signed by patient himself, a consent by a family member will be sought. As soon as possible, the patient will be informed and asked to sign a consent for continuing of study;
* Hemodynamic stability of patient during 1 hour without change in norepinephrine dosage;
* Treatment with noradrenaline for less than 48 hours.

Exclusion Criteria:

* Need of noradrenaline > 3 mg/h;
* Treatment with dobutamine;
* Personal history of severe asthma;
* Personal history of severe chronic obstructive pulmonary disease;
* Personal history of pulmonary hypertension;
* Personal history of second degree or third degree atrioventricular block without pacemaker;
* Personal history of sinoatrial block without pacemaker;
* Chronic heart failure with ejection fraction < 40%;
* Severe atrioventricular nodal bradycardia (heart rate < 70 bpm);
* Mean arterial pressure < 65 mm Hg;
* Hypersensitivity to esmolol;
* Prinzmetal angina;
* Pheochromocytoma without treatment;
* Pregnancy woman;
* Breastfeeding woman;
* Peripheral arterial disease;
* Patient with pacemaker;
* Chronic treatment with a beta blocker;
* Concomitant treatment with bepridil, diltiazem, verapamil, amiodarone, propafenone, Class Ia antiarrythmics (hydroquinidine, disopyramide) or baclofen;
* Patient < 18 years;
* Patient under the care of a guardian;
* Therapeutic futility;
* Lack of medical insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of hemodynamic parameters between 3 groups | 24 hours
  3 groups: GC, G10 and G20.
  The hemodynamic tolerance will be considered as satisfactory if the variation of MAP and cardiac output induced by esmolol does not exceed 15% of baseline (H0).
Immunomodulatory effect | 24 hours
  Immunomodulatory effect of esmolol will be evaluated notably by the ratio of IL6 / IL10.
  The decrease of this ratio in comparison with the value at baseline (H0) will be considered as an indicator of esmolol efficacy as immunomodulator.

SECONDARY OUTCOMES:
Comparison of number and severity of organ failures, between the 3 groups | 28 days
  3 groups will be evaluated by SOFA score.
Comparison of autonomic nervous system activity between the 3 groups | 24 hours
  Power spectrum analysis of heart rate variability.
Comparison of mortality in the 3 groups | 28 days
Comparison in the 3 groups of the correlations between the biomarkers and the hemodynamic data | 24 hours
  The biomarkers in plasma levels: cortisol, catecholamine, proinflammatory cytokines and anti-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Djillali ANNANE, MD, PhD, Principal Investigator — ICU, Hôpital Raymond Poincaré, 92380 Garches, France
Locations (1):
- ICU, Hôpital Raymond Poincaré, Garches, Haute Des Seine, France